CLINICAL TRIAL: NCT03828422
Title: Arterial Function and Atherosclerosis in Patients With JAK2 V167F Positive Essential Thrombocythemia
Brief Title: Arterial Function and Atherosclerosis in Essential Thrombocythemia
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Ales Blinc, Ales Blinc, MD, PhD, Head, Dept of Vascular Diseases, University Medical Centre Ljubljana
Other Study IDs: TP20180038
Record Dates: First submitted 2019-01-23; First posted 2019-02-04 (Actual); Results first posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Atherosclerosis
Keywords: essential thrombocythaemia; JAK2 V617F mutation burden; preclinical atherosclerosis; arterial stiffness; endothelial function; coronary artery calcium score
MeSH Terms: conditions — Atherosclerosis; Thrombocythemia, Essential | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The ipsogen JAK2 MutaQuant Kit, Qiagen (ZDA) (Ref: No. 673523) will be used for the detection and quantification of JAK2 V617F/G1849T allele in genomic DNA extracted from peripheral blood of patients and also control subjects. A SNP specific primer that selectively amplifies JAK2 V617F allele will be used with a real-time qPCR instrument which accurately quantifies the PCR products.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with essential thrombocythemia: * essential thrombocythemia with JAK2 V617F positive mutation
  * patients from the Department of Haematology at University Medical Centre Ljubljana, Slovenia, who were diagnosed with JAK2 V617F positive ET between 2011 and 2014
  * no personal history of clinically manifest atherosclerotic vascular disease (myocardial infarction, angina pectoris, peripheral arterial disease, aortic disease, transient ischemic attack or ischemic stroke)
  * all signed the informed consent
  * examined twice, the first time in the years 2014-2015 and for the second time in the years 2018-2019
  * blood for laboratory tests
  * imaging and functional examination: ultrasound examination, EndoPat plethysmography, coronary artery calcium scanning
  Interventions: Diagnostic Test: imaging
- control group: * the control group is selected among healthy employees of the University Medical Centre Ljubljana and their relatives
  * they are matched with the patient group for age and sex distribution and classical risk factors for cardiovascular disease
  * no personal history of clinically manifest atherosclerotic vascular disease (myocardial infarction, angina pectoris, peripheral arterial disease, aortic disease, transient ischemic attack or ischemic stroke)
  * all signed the informed consent
  * blood for laboratory tests
  * examined twice, the first time in the years 2014-2015 and for the second time the in years 2018-2019
  * imaging and functional examination: ultrasound examination, EndoPat plethysmography, coronary artery calcium scanning
  Interventions: Diagnostic Test: imaging

INTERVENTIONS:
Diagnostic Test: imaging
  Other Names: EndoPat plethysmography; coronary artery calcium scanning; blood laboratory tests; ultrasound examination

SUMMARY:
The aim of the study is to examine (a) whether patients with JAK2 V617F positive ET in comparison to age-and sex-matched, apparently healthy control subjects show more advanced progression of arterial stiffness, pulse-wave velocity and coronary calcium score in a 4 year observation period, and (b) whether the burden of JAK2 V617F mutation correlates with the measured vascular parameters. All subjects will be examined twice. The first visit already took place between the years 2014 - 2015 and the second visit will take place between 2018-2019. All participants will have signed their informed consent before entering the study. Each visit will consist of completing a structured questionnaire (on personal and family medical history, risk factors for CVD and medication), physical examination, donating a blood sample for laboratory tests and undergoing carotid ultrasound and coronary calcium measurement oft the extent of coronary artery calcification. At the first and the second examination the JAK2 V617F allele burden, i.e. the percentage of mutated alleles, will be determined from genomic DNA in peripheral blood.

DETAILED DESCRIPTION:
1. Patients and control subjects

   Patients are selected from the database of the Department of Haematology at University Medical Centre Ljubljana, Slovenia, who were diagnosed with JAK2 V617F positive ET between 2011 and 2014. There were 124 JAK2 positive ET patients, among those 61 did not have a personal history of clinically manifest atherosclerotic vascular disease (myocardial infarction, angina pectoris, peripheral arterial disease, aortic disease, transient ischemic attack or ischemic stroke). 40 patients (14 male and 26 female) with JAK2 V617F positive ET without clinically apparent cardiovascular disease signed the informed consent and were enrolled in the study in 2014 - 2015 for the first examination and 36 (12 male and 24 female) of them are expected to participate also in 2018-19.

   The control group is selected among healthy employees of the University Medical Centre Ljubljana and their relatives. It is matched with the patient group for age and sex distribution and classical risk factors for cardiovascular disease. 42 individuals (16 male and 26 female) participated in the first examination and at least 38 (14 male and 24 female) subjects are expected to paticipate in the second examination.
2. Baseline measurements

   Each participant will complete a questionnaire about family history of cardiovascular diseases, personal medical history, smoking status and medications. A physical examination will be performed, including measurements of height, weight, waist circumference, systolic and diastolic blood pressure. Blood will be sampled for laboratory analysis of complete blood cell count, electrolytes, serum lipids, liver function tests, urea, creatinine, and inflammatory markers.

   The 10-year risk of coronary heart disease (CHD) and general cardiovascular disease (CVD) will be calculated using the Framingham risk equation.
3. JAK2 V617F/G1849T allele burden

   The ipsogen JAK2 MutaQuant Kit, Qiagen (ZDA) (Ref: No. 673523) will be used for the detection and quantification of JAK2 V617F/G1849T allele in genomic DNA extracted from peripheral blood of patients and also control subjects. A SNP specific primer selectively amplifies the JAK2 V617F allele which is detected with a real-time qPCR instrument that quantifies the PCR products. The JAK2 V617F allele burden will be calculated and expressed as the percentage of JAK2 V617F mutated alleles throughout the whole JAK2 record. Analysis will be done done in laboratory of the Department of Haematology at University Medical Centre Ljubljana for all samples.
4. Carotid Artery Ultrasound Examination

   For examination of the extracranial carotid arteries an ultrasound machine Aloka Prosound α7 (Hitachi Aloka Medical, Ltd., Japan) will be used with a linear vascular probe working at a frequency of 5-13 MHz. The common, internal and external carotid arteries on both sided will be examined. At each examination, the measurements will be done twice and their average values will be calculated. The ultrasound examination will be done by the same ultrasonographer at both visits of all participants.

   The intima-media thickness will be measured 2 cm proximal to the bulb of common carotid artery on both sides. Screening of the extracranial carotid arteries for atherosclerotic plaques will be performed, with a plaque definition of a focal lesion, exceeding the intima-media thickness for at least 50% or reaching an absolute thickness of at least 1.5 mm in two orthogonal projections. Scoring of atherosclerotic plaques is done according to the methodology from the Rotterdam Study. The presence of at least one plaque in each segment of the extracranial carotid arterial bed, (divided into the common carotid artery and the bulb, the internal carotid artery and the external carotid artery) on either sides is scored 1 point. Thus, the carotid plaque score ranges from 0 (absence of plaques) to 6 (plaques present in all segments on both sides).

   Echo-tracking of the common carotid artery will be used to assess arterial stiffness expressed by the β-stiffness index and the pulse wave velocity. Measurements will be done at the common carotid artery 2 cm proximal to the bulb on both sides. The β-stiffness index will be calculated as: β = ln (P_max / P_min) / [(D_max - D_min / D_min)], where P_max = the systolic blood pressure, P_min = the diastolic pressure; D_max = the maximum arterial diameter and D_min = the minimal arterial diameter. Pulse wave velocity (PWV) will be calculated as: PWV = √ ((β x P_min) / 2ρ)); ρ = 1050 kg/m³.
5. Assessment of Endothelial Function of the Digital Arteries

   Endothelial function of the digital arteries will be measured by digital plethymography with EndoPat 2000, Itamar Medical REF, Caesarea, Israel, Software Version 3.3.x and expressed as the Reactive Hyperaemia Index (RHI) and the Augmentation Index (AI). Changes in arterial tone are elicited by creating a downstream hyperemic response induced by a standard 5-minute occlusion of the brachial artery (using a blood pressure cuff, inflated to 60 mmHg above the arterial blood pressure). When the cuff is released, the surge of blood flow causes endothelium-dependent flow mediated dilatation (FMD) which is manifested as reactive hyperemia. A post-occlusion to pre-occlusion ratio is calculated by EndoPAT software and the and A) are determined. The results are normalized to a heart rate of 75/min.
6. Measurement of the Coronary Artery Calcium Burden

   The calcium burden of coronary arteries is measured with a Biograph M 128-row PET-CT scanner (Siemens, Erlangen, Germany). Scanning is done from the base to the apex of the heart. A non-contrast protocol with sequential prospective ECG triggering is used. The rotation time is 0.33 sec, with a tube voltage of 120 kV, CARE Dose 4D and slice thickness 3 mm, with no slice overlap. Post-processing is done on the Syngo Leonardo workstation. The coronary calcium burden is expressed as the Agatston score. Evaluation of the dataset of every study subject is done three times and the average value is used for further analysis.
7. Statistical analysis

All sets of data will be tested for normality of distribution using the normal-quintile plot, calculating the correlation coefficient and checking it for the critical value that would warrant rejection of normal distribution with an α-error probability of 0.05.

Normally distributed data will be presented as mean and standard deviation, while non-normally distributed data will be presented as median and range between the 1st and 3rd quartile.

Differences between subjects with ET and control subjects at the first and second examination will be tested by the chi-square test for discrete variables, for normally distributed continuous variables by the paired Student's t-test for independent samples, and for non-normally distributed continuous variables by the Mann-Whitney test for independent samples. P-values of < 0.05 will be considered significant with a correction for multiple comparisons.

Changes in vascular function and morphology in the 4-year observation period will be compared between the two groups by the log rank test. P-values of < 0.05 will be considered significant.

The association between the parameters of vascular function / morphology and the JAK2 V617F allele burden will be assessed by the Pearson correlation coefficient.

ELIGIBILITY:
Inclusion Criteria:

* patients with JAK2 V617F positive essential thrombocythemia
* age-and sex-matched apparently healthy control subjects

Exclusion Criteria:

* personal history of any atherosclerotic vascular disease (myocardial infarction, angina pectoris, peripheral arterial disease, aortic disease, transient ischemic attack or ischemic stroke)
* chronic kidney disease stage 3 and above
* known cancer
* chronic inflammatory disease
* autoimmune disease
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Expected patient group: 40 patients (14 male and 26 female) with JAK2 V617F positive ET without clinically apparent cardiovascular disease. Average age 55,05 (13,48); ITM 25,22 (3,65); systolic blood pressure 138 (124-150) mmHg; diastolic blood pressure 81 (74-85) mmHg; Framingham risk score for CHD 6,84%.
  Expected control group: 42 individuals (16 male and 26 female) who were age and sex matched with the patient group. Average age 59,16 (12,03); ITM 27,27 (4,64); systolic blood pressure 132 (125-141) mmHg; diastolic blood pressure 81 (76-86) mmHg; Framingham risk score for CHD 7,20%.
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2021-08 (Actual); Study Completion 2021-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ales Blinc, MD, Study Director — University Medical Centre Ljubljana

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Vrtovec M, Anzic A, Zupan IP, Zaletel K, Blinc A. Carotid Artery Stiffness, Digital Endothelial Function, and Coronary Calcium in Patients with Essential Thrombocytosis, Free of Overt Atherosclerotic Disease. Radiol Oncol. 2017 Jan 14;51(2):203-210. doi: 10.1515/raon-2017-0006. eCollection 2017 Jun. PMID 28740456
- [Result] Anzic Drofenik A, Vrtovec M, Bozic Mijovski M, Sever M, Preloznik Zupan I, Kejzar N, Blinc A. Progression of coronary calcium burden and carotid stiffness in patients with essential thrombocythemia associated with JAK2 V617F mutation. Atherosclerosis. 2020 Mar;296:25-31. doi: 10.1016/j.atherosclerosis.2020.01.001. Epub 2020 Jan 11. PMID 32005002

RESULTS

PARTICIPANT FLOW:
Recruitment Details: a single tertiary medical centre
Pre-assignment Details: had documented or clinically suspected atherosclerotic vascular disease
Groups:
- Patients With Essential Thrombocythemia: * essential thrombocythemia with JAK2 V617F positive mutation
  * patients from the Department of Haematology at University Medical Centre Ljubljana, Slovenia, who were diagnosed with JAK2 V617F positive ET between 2011 and 2014
  * no personal history of clinically manifest atherosclerotic vascular disease (myocardial infarction, angina pectoris, peripheral arterial disease, aortic disease, transient ischemic attack or ischemic stroke)
  * all signed the informed consent
  * examined twice, the first time in the years 2014-2015 and for the second time in the years 2018-2019
  * blood for laboratory tests
  * imaging and functional examination: ultrasound examination, EndoPat plethysmography, coronary artery calcium scanning
  imaging
- Control Group: * the control group is selected among healthy employees of the University Medical Centre Ljubljana and their relatives
  * they are matched with the patient group for age and sex distribution and classical risk factors for cardiovascular disease
  * no personal history of clinically manifest atherosclerotic vascular disease (myocardial infarction, angina pectoris, peripheral arterial disease, aortic disease, transient ischemic attack or ischemic stroke)
  * all signed the informed consent
  * blood for laboratory tests
  * examined twice, the first time in the years 2014-2015 and for the second time the in years 2018-2019
  * imaging and functional examination: ultrasound examination, EndoPat plethysmography, coronary artery calcium scanning
  imaging
Period: Overall Study
Arm/Group | Patients With Essential Thrombocythemia | Control Group
Started | 40 | 42
Completed | 36 | 38
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Population: 4 participants did not particiapete at the second visit
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients With Essential Thrombocythemia | Control Group | Total
Number analyzed (Participants) | 36 | 38 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (13) | 59 (12) | 57 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 12 | 14 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Slovenia | 36 | 38 | 74

OUTCOME MEASURES:

1. Primary Outcome: Carotid Artery Stiffness (Expressed by Beta-stiffness Index ) in JAK2 V617F Positive ET Patients in Comparison to Healthy Control Subjects in a 4-year Period (From Baseline to Year 4).
Description: 4-year change carotid artery in Beta-stiffness Index measured in JAK2 V617F positive ET patients in comparison to healthy control subjects. All measurements were performed by echo-tracking ultrasound of the common carotid artery.
  Echo-tracking of the common carotid artery wall was used to assess arterial stiffness expressed by the β-stiffness index. Measurement swere done at the common carotid artery 2 cm proximal to the bulb on both sides. The β-stiffness index was calculated as: β = ln (P_max / P_min) / [(D_max - D_min / D_min)] (P_max = the systolic blood pressure, P_min = the diastolic pressure; D_max = the maximum arterial diameter and D_min = the minimal arterial diameter). In the adult population, the values of β range from 4 - 10 and increase with age. A larger value of β means increased arterial stiffness, i.e., a worse outcome.
Time Frame: From Baseline (in 2014-2015) to Year 4 (in 2018-2019)
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Patients With Essential Thrombocythemia | Control Group
Number analyzed (Participants) | 36 | 38
index | 1.95 (2.18) | 0.22 (1.99)

2. Primary Outcome: Carotid Artery Stiffness (Expressed by the Pulse Wave Velocity) in JAK2 V617F Positive ET Patients in Comparison to Healthy Control Subjects in a 4-year Period (From Baseline to Year 4).
Description: 4-year change in carotid artery pulse wave velocity (PWV) measured in JAK2 V617F positive ET patients in comparison to healthy control subjects. All measurements were performed by echo-tracking ultrasound of the common carotid artery.
  Measurements were done at the common carotid artery 2 cm proximal to the bulb on both sides. PWV was calculated from the beta stiffness index (β, for description see above), as follows:
  PWV = √ ((β x P_min) / 2ρ)); ρ = 1050 kg/m³. PWV increases with arterial stiffness, a larger value means a worse outcome. PWV in adults ranges from 3 m/s to 12 m/s; values are strongly age dependent.
Time Frame: From Baseline (in 2014-2015) to Year 4 (in 2018-2019)
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Patients With Essential Thrombocythemia | Control Group
Number analyzed (Participants) | 36 | 38
m/s | 0.72 (0.92) | 0.08 (0.72)

3. Primary Outcome: Change of Carotid Artery Plaque Score in JAK2 V617F Positive ET Patients in Comparison to Healthy Control Subjects in a 4-year Period.
Description: Change in carotid plaque score (i.e., the number of carotid artery segments with detected plaques, reported on a scale from 0-6) in a 4 year observation period.
  A carotid plaque score 0 means that the common carotid, internal carotid and exteranal carotid artery on both sides are free from plaques. A score of 6 means that the common carotid, internal carotid and external carotid artery on both sides have plaques detected by ultrasound.
Time Frame: From Baseline (in 2014-2015) to Year 4 (in 2018-2019)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Patients With Essential Thrombocythemia | Control Group
Number analyzed (Participants) | 36 | 38
score on a scale | 0 [0 to 0] | 0 [0 to 0]

4. Primary Outcome: Change of Coronary Calcium Burden in JAK2 V617F Positive ET Patients in Comparison to Healthy Control Subjects in a 4-year Period.
Description: Change in the Agatston coronary artery calcium score in a 4 year observation period.
  Agatston score denotes the number of coronary artery calcifications weighted for the intensity of calcification.
  Grading of coronary artery disease (CAD) based od Agatston score goes as follows: no CAD = score 0, minimal CAD = score 1-10, mild CAD = score 11-100, moderate CAD = score 101-400, svere CAD = score > 400.
Time Frame: From Baseline (in 2014-2015) to Year 4 (in 2018-2019)
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Patients With Essential Thrombocythemia | Control Group
Number analyzed (Participants) | 36 | 38
units on a scale | 0 [0 to 15.85] | 1.6 [0 to 14.10]

5. Primary Outcome: Change of Digital Endothelial Function, Expressed as Reactive Hyperemia Index and Augmentation Index (AI), in JAK2 V617F Positive ET Patients in Comparison to Healthy Control Subjects in a 4-year Period.
Description: 4-year change in Reactive Hyperemia Index (RHI) and 4-year change Augmentation Index (AI).
  RHI was calculated by the formula:
  RHI = (A/B) / (C/D) where A is the post-occlusion pulse wave amplitude (PWA) of the occluded hand, B the baseline PWA of the occluded hand, C the post-occlusion PWA of the contralateral hand, and D the baseline PWA of the contralateral hand. A higher RHI means better endothelial function (= good outcome). RHI in patients ranges from1-3. Arbitrarily, normal RHI is defined as => 1.67, and abnormal RHI as RHI =< 1.66.
  The AI was determined from the shape of the arterial pulse wave by the EndoPAT 2000 software which distinguished between the primary pulse wave (P1) and the reflected pulse wave (P2) by the formula: AI = ((P2-P1)/P1) x 100. The results were normalized to a heart rate of 75/min. A higher AI means greater arterial stiffness (= bad outcome). AI >0.4 is abnormal.
Time Frame: From Baseline (in 2014-2015) to Year 4 (in 2018-2019)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients With Essential Thrombocythemia | Control Group
Number analyzed (Participants) | 36 | 38
units on a scale
  Reactive Hyperemia Index (RHI) | -0.02 (0.77) | -0.26 (0.89)
  Augmentation Index (AI) | 3.56 (16.88) | 0.46 (20.19)

6. Primary Outcome: The JAK2 V617F Mutation Burden in Patients With JAK2 V617F Positive ET.
Description: Change in JAK2 V617F mutation burden in the 4-year observation period. Ipsogen JAK2 MutaQuant Kit, Qiagen (USA) was used for the detection of JAK2 V617F mutation and quantification of its burden in genomic DNA, which was extracted from granulocytes in peripheral blood. Real-time quantitative polymerase chain reaction (qPCR) was used with double-dye oligonucleotide hydrolysis principle. The JAK2 V617F burden was defined as the percentage of JAK2 V617F mutated alleles in total genomic DNA.
Time Frame: At baseline (in 2014- 2015) and at the second visit (in 2018-2019)
Population: The control group was not included in the comparison because they lack JAK2 V617F mutation as they are healthy subjects with no mutation. We examine the association between mutation burden (where the mutation is necessary) and coronary calcium burden.
Measure: Median (Inter-Quartile Range); unit: percentage of mutant allele
Arm/Group | Patients With Essential Thrombocythemia
Number analyzed (Participants) | 36
percentage of mutant allele
  JAK2 V617F mutation burden at baseline | 29.95 [7.32 to 43.33]
  JAK2 V617F mutation burden at the second visit | 11.60 [0 to 26.63]

ADVERSE EVENTS:
Time Frame: From Baseline (in 2014- 2015) to Year 4 (2018-2019)
Description: There were no adverse events.
Arm/Group | Patients With Essential Thrombocythemia | Control Group
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/38
Other Adverse Events (participants affected / at risk) | 0/36 | 0/38

LIMITATIONS AND CAVEATS:
* the relatively small number of participants (patients were recruited from a single tertiary medical centre)
* the subjects were not examined at precisely the same time interval between both visit

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-26): https://cdn.clinicaltrials.gov/large-docs/22/NCT03828422/Prot_SAP_000.pdf